CLINICAL TRIAL: NCT00182078
Title: A Study of Sertraline to Prevent PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Frederick J. Stoddard, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SHC Grant No. 8840; SHC Grant No. 8840 (Other Grant/Funding Number: Shriners Hospitals for Children); Protocol #:2002P001521; MGH (Other: Partners Human Research Committee)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: sertraline; children; adolescents; posttraumatic stress disorder; depression; prevention; burns; injuries
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Burns; Wounds and Injuries | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo was administered on a flexible fixed schedule and tapered at 12 weeks.
  Interventions: Drug: Placebo
- Sertraline (Experimental): Sertraline was administered on a flexible fixed schedule beginning at 25 mg/day and increasing as high as 150 mg/day. At week 12, the medication was tapered at a rate of 25 mg every 3 days until it was discontinued.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Placebo — The placebo was administered for 24 weeks on a flexible fixed schedule beginning at 25mg per day, and increasing as high as 150 mg/day. Both groups received the assigned medication and dose over a 24-week period. At Week 12, the placebo was tapered at a rate of 25mg every 3 days until it was discontinued.
  Arms: Placebo
Drug: Sertraline — The drugs were administered for 24 weeks on a flexible fixed schedule beginning at 25mg per day, and increasing as high as 150 mg/day. Both groups received the assigned medication and dose over a 24-week period. At Week 12, the medication was tapered at a rate of 25mg every 3 days until it was discontinued.
  Other Names: Zoloft
  Arms: Sertraline

SUMMARY:
The broad, long-term objectives of this proposal are to prevent the emergence of posttraumatic stress and depressive symptoms in children admitted for an acute burn, reconstructive surgery, or non-burn injury. This study is investigating the early use of a medication in the prevention of posttraumatic stress disorder and depression. Specific Aims 1 and 2: To assess the efficacy of sertraline to prevent the development of (Aim 1)posttraumatic stress disorder and (Aim 2)depression in children aged 6-20, after burn or non-burn injury or after reconstructive surgery. Hypotheses 1 and 2: Administration of sertraline after an acute burn or non-burn injury, or after reconstructive surgery will lead to greater reduction in post-traumatic and depressive symptoms over 12 and 24 weeks, compared with placebo.

This study is completing the evaluation of 90 children and adolescents, aged 6-20 years. It is comparing 60 subjects receiving sertraline with 30 placebo control subjects matched for age, severity of injury, and type of hospitalization (acute vs. reconstructive). Children and families are evaluated for the presence of acute stress symptoms. Children are reassessed in a double-blind placebo-controlled design, with evaluations at Baseline, Week 2, Week 4, Week 8, Week 12, and Week 24. In addition, there is weekly monitoring for the first 14 weeks of the study and again at 18 weeks (the midpoint of the study). At each reassessment, information is collected on the child's compliance with the study medication, the parents' assessment of the child's functioning, and the child's self-report of posttraumatic and depressive symptomatology. The main outcome variable used in this study is the child's posttraumatic symptoms.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

1. SPECIFIC AIM 1: To assess the efficacy of sertraline in preventing posttraumatic stress disorder in children aged 6-20 after a burn, injury or reconstructive surgery following a burn injury.
2. SPECIFIC AIM 2: To assess the efficacy of sertraline in preventing co-morbid depression in children aged 6-20 after a burn, injury or reconstructive surgery following a burn injury.

BACKGROUND AND SIGNIFICANCE Prevention of posttraumatic stress symptoms is a priority in psychiatric practice today. This is the first controlled study of any medication to prevent posttraumatic stress disorder (PTSD) in children and adolescents. The purpose of the study is to use sertraline to prevent PTSD and co-morbid depression from developing in 6-20 year old children hospitalized with a burn, injury, or reconstructive surgery following a burn injury. If this intervention is successful, it will help to prevent psychiatric and developmental disorders in injured children as well as those who undergo reconstructive procedures. While we have found no studies that have investigated the efficacy of sertraline in treating PTSD in children and adolescents, research indicates that sertraline is effective in treating other anxiety disorders and depression in children and adolescents. Research also indicates that sertraline is effective in treating PTSD in adults.

RECRUITMENT PROCEDURES Families of children aged 6-20 admitted with an acute burn or for reconstructive surgery are contacted by study staff within 3 days of admission or when medically stable, and asked to participate in the study. In addition, 6-17 year old patients admitted for an injury are asked to participate.

CONSENT PROCEDURES: A licensed physician investigator explains the nature of the study and requests consent from the child's primary caregiver or legal guardian as soon as possible after hospital admission. Once consent is given, the research coordinator obtains the baseline data.

Ninety children will be enrolled in the study. These children must a) be a burn patient between the ages of 6 and 20 or an injured patient between the ages of 6-17, b) have responded to the burn, injury, or surgery with fear, helplessness, or horror, and c) be proficient in English or Spanish. If a child has no memory of the injury, currently uses antidepressants, or has a known sensitivity to sertraline, diagnosis of Bipolar disorder, diagnosis of PTSD, mental retardation, Traumatic Brain Injury, or a new onset of seizures or marked worsening of a seizure disorder, he/she will not be included in the study.

STUDY PROCEDURES After the child is enrolled, he/she is randomly assigned to receive either sertraline or placebo. Neither the family nor the investigator will know which group the child is assigned to. If at any time this information becomes medically necessary, it will be made available to the child's doctor.

The child takes the study medication every day for 12 weeks. If the child is in the sertraline group, the dose of medication may be increased gradually until a satisfactory response is achieved. If the child is in the placebo group, he/she may receive sertraline after 12 weeks if clinically indicated. After 12 weeks, the medication or placebo will be tapered at a rate of 25 mg every three days.

All children and families are assessed at six points: Early in their acute hospitalization (Baseline), at again at weeks 2, 4, 8, 12, and 24. The baseline and follow-up assessments of 8, 12, and 24 weeks include child and parent interviews. During each assessment, the child and parent complete several questionnaires examining how the child is functioning. Check up assessments are completed as recommended by the FDA. The assessments take place in the hospital, at home, or by the telephone after the child had been discharged.

EQUITABLE SELECTION OF SUBJECTS Proficiency in English or Spanish is needed in order to be included in the study as the study instruments are not validated for non-English and non-Spanish speaking populations.

PRIVACY AND CONFIDENTIALITY Parents/guardians are informed that the information gathered in the study is confidential and will not adversely affect their child's treatment in any way. The child is assigned a research identification number and this number, not their name, will be placed on the study questionnaires. The document that matches name with identification number is kept in a locked cabinet that is accessible only to study staff. The data stored in the computer is password protected and computer access is limited to study staff. All interview and questionnaire data is kept in a locked cabinet. Families are also told prior to entering the study that certain information (i.e., suspicions of child abuse or neglect) cannot be confidential.

EXPECTED BENEFITS The child's psychiatric symptoms may potentially decrease as a result of taking sertraline. If sertraline is found to prevent PTSD, the patient and other children will benefit from its use. In addition, the child may benefit from on-going psychological follow-up over the course of 24-weeks. At the conclusion of the study, the family has an opportunity to meet with one of the investigators and discuss the results of the evaluation.

Potential benefits to society: This study may be helpful in scientifically understanding the effect of sertraline on children's psychological and physiological responses to stress. It may be satisfying to families to learn that they are contributing to a body of knowledge that may help children/adolescents who are burned or injured in other ways. It is our hope that sertraline will help to prevent the debilitating symptoms of PTSD among burned and injured children and adolescents. Because PTSD can have long-lasting impacts both on the developing brain as well as on functional development, the successful prevention of the development of these symptoms would have far-reaching beneficial implications for children suffering burn injuries, as well as those suffering other forms of physical and psychological trauma.

FORESEEABLE RISKS AND DISCOMFORTS Sertraline has been shown to be well tolerated by both children and adolescents. Its side effects may include nausea, headache, stomach distress, diarrhea, dry mouth, insomnia, sexual dysfunction, sleepiness, dizziness, tremor, and fatigue. Most side effects appear early in treatment, and for about 10% of people it leads to stopping treatment. After tapering off the sertraline, these side effects will gradually stop also.

Because drugs that affect the nervous system can affect judgment, thinking or coordination, subjects will be warned to be cautious about operating hazardous machinery, including automobiles, until there is reasonable certainty that subjects are not affected adversely by this drug treatment.

We ask subjects to avoid alcoholic beverages during this study. It is possible that the combination of alcohol and medication may cause unknown side effects. Use of illegal drugs is prohibited.

Stopping the medication abruptly may be dangerous, hence, we inform the subjects that a gradual decrease in medication dose will be necessary for medication discontinuation. The risks of suddenly stopping the mediation include the possibility of nausea, malaise, muscle aches, headaches, mood changes, and unusual sensations (numbness and tingling). Subjects should contact the investigator before discontinuing the medication.

If the side effects of the medication are too uncomfortable and remain so, the sertraline may be decreased, or tapered and stopped, and alternative treatments will be offered, including counseling and/or alternative medications. If a subject remains distressed, doctors are available to help for as long as the subject is in the hospital. If, after the subject leaves the hospital and needs more treatment, the study doctors will refer him/her to a mental health professional in the community. If during this study the subject becomes distressed, he/she will have the opportunity to call and be evaluated by study staff.

Individuals with bipolar disorder (manic-depressive illness) cannot participate in the study because of the risk of inducing mania or hypomania with anti-depressants.

Due to potential for fatal interaction, subjects should avoid taking monoamine oxidase inhibitors (MAOIs) within at least 30 days of taking sertraline, and should avoid starting MAOI treatment until at least 30 days after discontinuation of treatment with sertraline.

Subjects may experience an allergic reaction to sertraline, or placebo ingredients. If a subject experiences allergy symptoms such as rash, hives or itching, he/she should notify their doctor immediately. Untreated allergy symptoms can lead to a medical emergency. Since this is a research study and the treatments or procedures are relatively new, there may be additional risks or side effects that we do not know about at this time, but which might occur during the study or later. Subjects will be informed of any significant new information regarding sertraline that may affect their willingness to continue participation in the study. If subjects plan to take any drug other than the study medication or undergo any medical treatment, then we ask them to notify the study doctor before starting the drug or treatment. This applies to prescription drugs, over-the-counter drugs such as cough and cold remedies, antacids, investigational drugs/procedures, and sleeping medications. If surgery or a diagnostic procedure is planned, then the study doctor has to be notified before the procedure is performed.

Pregnant women and nursing mothers cannot participate in this study. It is important that subjects avoid pregnancy throughout this study because the use of any drug during pregnancy has the potential to harm the embryo or the fetus. We will instruct women of childbearing potential that they must reliably practice an approved form of birth control while participating in the study. If a subject does become pregnant, she must tell the study doctor immediately. Her participation in the study may end and she may need counseling for her pregnancy. If a subject becomes pregnant during the study or 15 days after her last dose of the medication and her pregnancy is carried to term, the investigator will ask her permission to follow the course of her pregnancy and delivery as well as the condition of her newborn. If a subject misses a period or thinks she might be pregnant during the study, she must notify her study doctor immediately so that she can be withdrawn from the study.

MINIMIZATION OF RISKS AND SAFETY MONITORING Source data is monitored by the co-investigators in the study. Safety and outcomes monitoring are conducted in accord with the rules and regulations of the Massachusetts General Hospital. Adverse events monitoring is conducted in accord with the policies and procedures of the Massachusetts General Hospital, and reported to the Human Research Committee of the Massachusetts General Hospital, in accord with Partners Human Research Committee Adverse Event Reporting Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Shriners Hospital or Massachusetts General Hospital for an acute burn, injury, or reconstructive surgery following a burn
* Between the ages of 6 - 20 years
* Recent experience of an acute burn, injury, or surgery meeting the Diagnostic and Statistical Manual(DSM-IV) A1 stressor criterion
* Child's response to the stressor meets Diagnostic and Statistical Manual(DSM-IV) A2 response criterion
* Proficiency in either English or Spanish

Exclusion Criteria:

* No memory of the injury
* Current use of an anti-depressant
* Known hypersensitivity to sertraline
* Diagnosis of Bipolar Disorder
* Diagnosis of PTSD
* Mental Retardation
* Traumatic Brain Injury
* New onset or marked worsening of a seizure disorder

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2002-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick J Stoddard, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Saxe GN, Stoddard F, Hall E, Chawla N, Lopez C, Sheridan R, King D, King L, Yehuda R. Pathways to PTSD, part I: Children with burns. Am J Psychiatry. 2005 Jul;162(7):1299-304. doi: 10.1176/appi.ajp.162.7.1299. PMID 15994712
- [Background] Stoddard FJ, Saxe G. Ten-year research review of physical injuries. J Am Acad Child Adolesc Psychiatry. 2001 Oct;40(10):1128-45. doi: 10.1097/00004583-200110000-00007. PMID 11589526
- [Background] Saxe G, Stoddard F, Courtney D, Cunningham K, Chawla N, Sheridan R, King D, King L. Relationship between acute morphine and the course of PTSD in children with burns. J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):915-21. doi: 10.1097/00004583-200108000-00013. PMID 11501691
- [Background] Stoddard FJ, Sheridan RL, Saxe GN, King BS, King BH, Chedekel DS, Schnitzer JJ, Martyn JA. Treatment of pain in acutely burned children. J Burn Care Rehabil. 2002 Mar-Apr;23(2):135-56. doi: 10.1097/00004630-200203000-00012. PMID 11882804
- [Background] Saxe G, Chawla N, Stoddard F, Kassam-Adams N, Courtney D, Cunningham K, Lopez C, Hall E, Sheridan R, King D, King L. Child Stress Disorders Checklist: a measure of ASD and PTSD in children. J Am Acad Child Adolesc Psychiatry. 2003 Aug;42(8):972-8. doi: 10.1097/01.CHI.0000046887.27264.F3. PMID 12874500
- [Background] Stoddard FJ, Todres ID. A new frontier: posttraumatic stress and its prevention, diagnosis, and treatment. Crit Care Med. 2001 Mar;29(3):687-8. doi: 10.1097/00003246-200103000-00050. No abstract available. PMID 11379543
- [Background] Stoddard FJ, Usher CT, Abrams AN. Psychopharmacology in pediatric critical care. Child Adolesc Psychiatr Clin N Am. 2006 Jul;15(3):611-55. doi: 10.1016/j.chc.2006.02.005. PMID 16797442
- [Result] Stoddard FJ Jr, Luthra R, Sorrentino EA, Saxe GN, Drake J, Chang Y, Levine JB, Chedekel DS, Sheridan RL. A randomized controlled trial of sertraline to prevent posttraumatic stress disorder in burned children. J Child Adolesc Psychopharmacol. 2011 Oct;21(5):469-77. doi: 10.1089/cap.2010.0133. PMID 22040192
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- See also: American Academy of Child and Adolescent Psychiatry — http://www.aacap.org/
- See also: American Psychiatric Association — http://www.psych.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants and their guardians were recruited from a major pediatric burn center for an acute burn or for reconstructive surgery for a burn.
Pre-assignment Details: One participant withdrew consent prior to starting the study medication.
Groups:
- Placebo - Received Placebo: The placebo was administered for 24 weeks on a flexible fixed schedule beginning at 25mg per day, and increasing as high as 150 mg/day. Both groups received the assigned medication and dose over a 24-week period. At Week 12, the placebo was tapered at a rate of 25mg every 3 days until it was discontinued.
- Sertraline - Received Study Medication: The drugs were administered for 24 weeks on a flexible fixed schedule beginning at 25mg per day, and increasing as high as 150 mg/day. Both groups received the assigned medication and dose over a 24-week period. At Week 12, the medication was tapered at a rate of 25mg every 3 days until it was discontinued.
Period: Overall Study
Arm/Group | Placebo - Received Placebo | Sertraline - Received Study Medication
Started | 9 | 17
Completed | 8 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was conducted with participants using available data. The different number participants who completed measures at the final time point is as follows: DICA-Parent (6 placebo, 15 sertraline); DICA-Child (6 placebo, 16 sertraline); and CDI (4 placebo, 16 sertraline).
Groups:
- Placebo: Placebo group who received no study medication.
- Sertraline: Sertraline group received study medication every day for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sertraline | Total
Number analyzed (Participants) | 9 | 17 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 17 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (3.5) | 12.3 (3.9) | 12.35 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 9 | 17 | 26

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Interview Schedule for Children and Adolescents (DICA) - Parent
Description: The DICA is a semi-structured interview, and was used to measure post Traumatic Stress Disorder (PTSD) symptoms in children. The DICA was administered to parents who were English-speaking. A minimum total score of 7 and a maximum total score of 18 is required to meet criteria for PTSD. A higher score is indicative of increased PTSD symptoms. Changes in scores from Baseline to Week 24 were examined.
Time Frame: Baseline to Week 24
Population: Intention to treat (ITT). Analysis was conducted on participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 6 | 15
units on a scale | -0.2 (2.6) | -4.0 (3.6)
Statistical Analysis 1: Comparison: Placebo vs Sertraline; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = 3.8, Standard Deviation 3.4

2. Secondary Outcome: The Child Depression Inventory (CDI)
Description: The CDI contains 27 items, and measures symptoms of depression in children and adolescents. The CDI ranges in score from 0-54, where higher scores are indicative of a greater number of symptoms. Changes in scores from Baseline to Week 12 were examined.
Time Frame: Baseline to Week 12
Population: Intention to treat (ITT). Analysis was conducted on participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 4 | 16
units on a scale | -7.5 (1.3) | -2.4 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Sertraline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 5.1, Standard Deviation 3.9

3. Primary Outcome: Diagnostic Interview for Children and Adolescents (DICA) - Child
Description: The DICA is a semi-structured interview, and was used to measure Post Traumatic Stress Disorder (PTSD) symptoms in children. The DICA was administered to children who were English-speaking. A minimum total score of 7 and a maximum total score of 18 is required to meet criteria for PTSD. A higher score is indicative of increased PTSD symptoms. Changes in scores from Baseline to Week 24 were examined.
Time Frame: Baseline to Week 24
Population: Intention to treat (ITT). Analysis was conducted on participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 6 | 16
units on a scale | -3.8 (3.5) | -4.7 (4.7)
Statistical Analysis 1: Comparison: Placebo vs Sertraline; Test type: Superiority or Other; p = 0.65, t-test, 2 sided; Mean Difference (Final Values) = 0.9, Standard Deviation 4.4

ADVERSE EVENTS:
Arm/Group | Placebo | Sertraline
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/17
Other Adverse Events (participants affected / at risk) | 0/9 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Sertraline (N=17)
Suicidal ideation. Tremors (Psychiatric disorders) | 0 (0) | 1 (1) — 1 subject in the sertraline arm was reported after discharge by his mother to have "tremors" and 1 incident of suicidal ideation(SI) when stressed with her. The tremors stopped after 1 week. No SI was present on evaluation, nor on followup.

LIMITATIONS AND CAVEATS:
One limitation of this study was the small sample size, due to the challenge of recruiting traumatized children and their parents for participation in a randomized controlled trial of a medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes